CLINICAL TRIAL: NCT03973905
Title: Effectiveness of Maternal Immunization With Boostrix at Preventing Pertussis Among Infants <2 Months Old in the United States: Analysis of a Dataset From a Case-control Study
Brief Title: Effectiveness of Maternal Immunization With Boostrix at Preventing Pertussis Among Infants <2 Months Old in the United States
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 210031
Record Dates: First submitted 2019-02-13; First posted 2019-06-04 (Actual); Results first posted 2020-07-07 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: Whooping Cough
Keywords: Whooping Cough; Boostrix; Tdap; effectiveness; pregnancy; infants
MeSH Terms: conditions — Whooping Cough

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- Pertussis Case Group: Infant subjects of at least 2 days old and less than (<) 2 months old, who met the pertussis diagnosis definition (laboratory confirmed pertussis, epidemiological linkage to a laboratory-confirmed case, clinically compatible illness), and who met the case infants inclusion criteria (resided in the catchment area on their cough onset date, were born in a hospital in their state of residence, had at least 37 weeks gestational age at birth, were neither adopted, nor in foster care and did not live in a residential care facility).
  This post-hoc analysis was limited to cases and controls whose mothers were either vaccinated with Boostrix or did not receive any Tdap vaccine. Cases with no remaining matched control were also excluded from the analysis and vice versa.
  Interventions: Other: Not applicable / dataset analysis
- Control Group: Infant subjects of at least 2 days old and less than (<) 2 months old, who did not have a pertussis diagnosis prior to the cough onset date and who met the inclusion criteria for control infants (were born on a hospital in their state of residence, were at least 37 weeks gestational age at birth, were neither adopted, nor in foster care, did not live in a residential care facility, were born at the same hospital as the case infant).
  This post-hoc analysis was limited to cases and controls whose mothers were either vaccinated with Boostrix or did not receive any Tdap vaccine. Cases with no remaining matched control were also excluded from the analysis and vice versa.
  Interventions: Other: Not applicable / dataset analysis

INTERVENTIONS:
Other: Not applicable / dataset analysis — Not applicable / dataset analysis

SUMMARY:
The purpose of this study is to estimate the effectiveness of maternal immunization with Boostrix at preventing pertussis in infants in the United States.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for case infants:

* Case infants were eligible for the enrolment if they:
* were at least 2 days old and < 2 months old on the cough onset date
* resided in the catchment area on their cough onset date
* were born in a hospital in their state of residence
* were ≥37 weeks' gestational age at birth
* were neither adopted nor in foster care
* did not live in a residential care facility

Inclusion criteria for control infants:

* Control infants were eligible for the enrolment if they:
* were at least 2 days old and <2 months old on the case infant's cough onset date
* were born in a hospital in their state of residence
* were ≥37 weeks' gestational age at birth
* were neither adopted nor in foster care
* did not live in a residential care facility
* were born at the same hospital as the case infant

did not have pertussis diagnosis prior to the cough onset date of the corresponding case infant

Exclusion Criteria:

* Infants (case and controls) whose mothers have received Adacel or mothers without brand information available, as well as controls who were matched to a case whose mother received Adacel or mothers without brand information available, will be excluded from the analysis of the effectiveness of vaccination with Boostrix.

Ages: 2 Days to 2 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Infant subjects, born to mothers exposed, or unexposed to Boostrix or any Tdap vaccination, coming from 6 emerging program network sites.
Sampling Method: Probability Sample
Enrollment: 290 (Actual)
Dates: Start 2019-02-15 (Actual); Primary Completion 2019-05-15 (Actual); Study Completion 2019-05-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Wavre, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Skoff TH, Blain AE, Watt J, Scherzinger K, McMahon M, Zansky SM, Kudish K, Cieslak PR, Lewis M, Shang N, Martin SW. Impact of the US Maternal Tetanus, Diphtheria, and Acellular Pertussis Vaccination Program on Preventing Pertussis in Infants <2 Months of Age: A Case-Control Evaluation. Clin Infect Dis. 2017 Nov 29;65(12):1977-1983. doi: 10.1093/cid/cix724. PMID 29028938

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The present analysis has been performed on the data set of a case-control study conducted in 6 US Emerging Infection Program Network states, either statewide (4 states) or in select counties (2 states) by Skoff et al., 2017.
Pre-assignment Details: The primary study was a case-control study evaluating the effectiveness of tetanus toxoid, reduced diphtheria toxoid, and acellular pertussis (Tdap) vaccines (Boostrix and Adacel) administered during pregnancy in preventing pertussis in infants.
Groups:
- Pertussis Case Group: Infant subjects of at least 2 days old and less than (<) 2 months old, who met the pertussis diagnosis definition (laboratory confirmed pertussis, epidemiological linkage to a laboratory-confirmed case, clinically compatible illness), and who met the case infants inclusion criteria (resided in the catchment area on their cough onset date, were born in a hospital in their state of residence, had at least 37 weeks gestational age at birth, were neither adopted, nor in foster care and did not live in a residential care facility) This post-hoc analysis was limited to cases and controls whose mothers were either vaccinated with Boostrix or did not receive any Tdap vaccine. Cases with no remaining matched control were also excluded from the analysis and vice versa.
- Control Group: Infant subjects of at least 2 days old and less than (<) 2 months old, who did not have a pertussis diagnosis prior to the cough onset date and who met the inclusion criteria for control infants (were born on a hospital in their state of residence, were at least 37 weeks gestational age at birth, were neither adopted, nor in foster care, did not live in a residential care facility, were born at the same hospital as the case infant) This post-hoc analysis was limited to cases and controls whose mothers were either vaccinated with Boostrix or did not receive any Tdap vaccine. Cases with no remaining matched control were also excluded from the analysis and vice versa.
Period: Overall Study
Arm/Group | Pertussis Case Group | Control Group
Started | 107 | 183
Completed | 107 | 183
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pertussis Case Group | Control Group | Total
Number analyzed (Participants) | 107 | 183 | 290
Age, Continuous [Mean (Standard Deviation); unit: Weeks]
  Infant's age (weeks) | 5.0 (1.9) | 4.8 (2.0) | 4.9 (2.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49 | 90 | 139
  Male | 58 | 93 | 151
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 88 | 140 | 228
  Black | 9 | 13 | 22
  Other-unspecified | 10 | 30 | 40

OUTCOME MEASURES:

1. Primary Outcome: Number of Pertussis Cases and Matched Controls Among Infants Born to Mothers Vaccinated With Boostrix Vaccine (During Third Trimester of Pregnancy) or Not Exposed to Any Tdap Vaccine During Pregnancy
Description: Vaccine effectiveness at preventing pertussis occurrence in infants < 2 months old is assessed by comparing the Boostrix immunization status during the third pregnancy trimester in mothers of infant pertussis cases and matched controls. The association between maternal Boostrix vaccination and pertussis in infants was analyzed using conditional logistic regression. The multivariate analysis was performed to obtain the adjusted values. Covariates that were statistically significant in the univariate analysis or considered as clinically significant were included in the multivariable conditional logistic regression model. Subjects with missing or unknown values, if any, for at least one of the risk factors were excluded from the model.
Time Frame: During the data collection period (from 1 January 2011 to 31 December 2014)
Population: The analysis includes cases and at least one matched control born from mothers either unvaccinated or vaccinated with Boostrix. Subjects with missing or unknown values, if any, for at least one of the risk factors were excluded from the model.
Measure: Count of Participants; unit: Participants
Arm/Group | Pertussis Case Group | Control Group
Number analyzed (Participants) | 106 | 180
Participants
  Unvaccinated | 72 | 112
  Vaccinated during third trimester | 5 | 17
Statistical Analysis 1: Comparison: Pertussis Case Group vs Control Group; To assess the effectiveness of maternal vaccination with Boostrix during third trimester of pregnancy (at least 14 days before delivery) at preventing pertussis in infants <2 months; Test type: Other; Vaccine Effectiveness = 65.26, 95% CI 2-sided [-64.93 to 92.68] — Vaccine Effectiveness (VE) was estimated as (1-odds ratio) × 100%. The Confidence Interval was calculated based on the conditional binomial distribution of cases in the exposed group and the total number of cases

2. Secondary Outcome: Number of Pertussis Cases and Matched Controls Among Infants Born to Mothers Vaccinated With Boostrix Vaccine (Before Pregnancy, During First or Second Trimester, After Pregnancy) or Not Exposed to Any Tdap Vaccine During Pregnancy
Description: Vaccine effectiveness at preventing pertussis occurrence in infants < 2 months old is assessed by comparing the Boostrix immunization status before pregnancy, during first or second pregnancy trimester, after pregnancy in mothers of infant pertussis cases and matched controls. The association between maternal Boostrix vaccination and pertussis in infants was analyzed using conditional logistic regression. The multivariate analysis was performed to obtain the adjusted values. Covariates that were statistically significant in the univariate analysis or considered as clinically significant were included in the multivariable conditional logistic regression model. Subjects with missing or unknown values, if any, for at least one of the risk factors were excluded from the model.
Time Frame: During the data collection period (from 1 January 2011 to 31 December 2014)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Pertussis Case Group | Control Group
Number analyzed (Participants) | 106 | 180
Participants
  Unvaccinated | 72 | 112
  Vaccinated, before pregnancy | 1 | 4
  Vaccinated, during first or second trimester | 1 | 6
  Vaccinated, after pregnancy | 27 | 41
Statistical Analysis 1: Comparison: Pertussis Case Group vs Control Group; To assess the effectiveness of maternal vaccination with Boostrix before pregnancy at preventing pertussis in infants <2 months; Test type: Other; Vaccine Effectiveness = 42.01, 95% CI 2-sided [-1071.80 to 97.13] — VE was estimated as (1-odds ratio) × 100%. The Confidence Interval was calculated based on the conditional binomial distribution of cases in the exposed group and the total number of cases
Statistical Analysis 2: Comparison: Pertussis Case Group vs Control Group; To assess the effectiveness of maternal vaccination with Boostrix during first or second trimester of pregnancy at preventing pertussis in infants <2 months; Test type: Other; Vaccine Effectiveness = 62.17, 95% CI 2-sided [-439.75 to 97.35] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: Pertussis Case Group vs Control Group; To assess the effectiveness of maternal vaccination with Boostrix after pregnancy at preventing pertussis in infants <2 months; Test type: Other; Vaccine Effectiveness = -12.89, 95% CI 2-sided [-166.37 to 52.16] — [estimate comment as in outcome 2, analysis 1]

3. Secondary Outcome: Number of Pertussis Cases and Matched Controls Among Infants Born to Mothers Vaccinated With Boostrix Vaccine (During First, Second or Third Trimester) or Not Exposed to Any Tdap Vaccine During Pregnancy
Description: Vaccine effectiveness at preventing pertussis occurrence in infants < 2 months old is assessed by comparing the Boostrix immunization status during pregnancy in mothers of infant pertussis cases and matched controls. The association between maternal Boostrix vaccination and pertussis in infants was analyzed using conditional logistic regression. The multivariate analysis was performed to obtain the adjusted values. Covariates that were statistically significant in the univariate analysis or considered as clinically significant were included in the multivariable conditional logistic regression model. Subjects with missing or unknown values, if any, for at least one of the risk factors were excluded from the model.
Time Frame: During the data collection period (from 1 January 2011 to 31 December 2014)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Pertussis Case Group | Control Group
Number analyzed (Participants) | 106 | 180
Participants
  Unvaccinated | 72 | 112
  Vaccinated, during pregnancy (Any trimester) | 6 | 23
Statistical Analysis 1: Comparison: Pertussis Case Group vs Control Group; To assess the effectiveness of maternal vaccination with Boostrix at any time during pregnancy at preventing pertussis in infants <2 months; Test type: Other; Vaccine Effectiveness = 64.79, 95% CI 2-sided [-57.51 to 92.13] — [estimate comment as in outcome 2, analysis 1]

4. Secondary Outcome: Number of Pertussis Cases Leading to Hospitalization and Matched Controls in Infants Born to Mothers Vaccinated With Boostrix (Before Pregnancy, During First or Second, Third Trimester, After Pregnancy) or Not Exposed to Any Tdap Vaccine During Pregnancy
Description: Vaccine effectiveness at preventing pertussis occurrence leading to hospitalization in infants < 2 months old is assessed by comparing the Boostrix immunization status before pregnancy, during first or second, third trimester, after pregnancy in mothers of infant pertussis cases and matched controls. The association between maternal Boostrix vaccination and pertussis in infants was analyzed using conditional logistic regression. The multivariate analysis was performed to obtain the adjusted values. Covariates that were statistically significant in the univariate analysis or considered as clinically significant were included in the multivariable conditional logistic regression model. Subjects with missing or unknown values, if any, for at least one of the risk factors were excluded from the model.
Time Frame: During the data collection period (from 1 January 2011 to 31 December 2014)
Population: The analysis includes cases leading to hospitalization and at least one matched control born from mothers either unvaccinated or vaccinated with Boostrix. Subjects with missing or unknown values, if any, for at least one of the risk factors were excluded from the model.
Measure: Count of Participants; unit: Participants
Arm/Group | Pertussis Case Group | Control Group
Number analyzed (Participants) | 69 | 121
Participants
  Unvaccinated | 49 | 78
  Vaccinated, before pregnancy | 1 | 2
  Vaccinated, during first or second trimester | 0 | 5
  Vaccinated, during third trimester | 3 | 11
  Vaccinated, after pregnancy | 16 | 25
Statistical Analysis 1: Comparison: Pertussis Case Group vs Control Group; [analysis description as in outcome 2, analysis 1]; Test type: Other; Vaccine Effectiveness = 17.65, 95% CI 2-sided [-12529.0 to 99.46] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Pertussis Case Group vs Control Group; To assess the effectiveness of maternal vaccination with Boostrix during third trimester of pregnancy at preventing pertussis in infants <2 months; Test type: Other; Vaccine Effectiveness = 85.01, 95% CI 2-sided [-13.91 to 98.03] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: Pertussis Case Group vs Control Group; [analysis description as in outcome 2, analysis 3]; Test type: Other; Vaccine Effectiveness = 37.64, 95% CI 2-sided [-87.40 to 79.25] — [estimate comment as in outcome 2, analysis 1]

ADVERSE EVENTS:
Description: All-Cause Mortality, Serious Adverse Events and Other Adverse Events were not collected/monitored in this observational study.
Arm/Group | Pertussis Case Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Due to the specificities of this project, developing both protocol and statistical analysis plan would have been redundant and of no added value. GSK therefore described the planned analysis in a detailed statistical analysis plan.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Statistical Analysis Plan (2019-03-08): https://cdn.clinicaltrials.gov/large-docs/05/NCT03973905/SAP_000.pdf
  • Study Protocol (2020-06-24): https://cdn.clinicaltrials.gov/large-docs/05/NCT03973905/Prot_001.pdf